CLINICAL TRIAL: NCT02637635
Title: Does Pre-treatment With Autologous Fat Transplantation Improve Results and Reduce Complication Rate After Breast Reconstruction With Implants? A Randomized Controlled Study
Brief Title: Does Autologous Fat Transplantation Improve Results and Reduce Complications in Breast Reconstruction With Implants?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Marie Wickman Chantereau, Adjunct professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCTLIP1
Record Dates: First submitted 2014-12-22; First posted 2015-12-22 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Breast Neoplasms
Keywords: Mammaplasty; Transplantation, Autologous; Mastectomy; Breast Implants; Radiotherapy, Adjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breast reconstruction with implant (Experimental): The patients will undergo breast reconstruction with an expander prosthesis.
  Interventions: Procedure: Expander prosthesis
- Autologous fat transplantation (Experimental): The patients will undergo lipofilling as a pre-treatment before they will undergo breast reconstruction with an expander prosthesis.
  Interventions: Procedure: Autologous fat transplantation; Procedure: Expander prosthesis

INTERVENTIONS:
Procedure: Autologous fat transplantation — 100 ml of autologous fat will be injected to the reconstruction area 3 month prior the breast reconstruction with expander prosthesis.
  Other Names: lipofilling; fat grafting; lipomodelling
  Arms: Autologous fat transplantation
Procedure: Expander prosthesis — breast reconstruction with expander prosthesis.
  Other Names: implant

SUMMARY:
The purpose of this study is to determine if autologous fat transplantation as a pre-treatment gives better results in breast reconstruction with implants after mastectomy and radiotherapy. One group is randomized to conventional reconstruction with implant and one to pre-treatment prior reconstruction with implant.

Our aims are:

1. To study whether lipofilling can decrease the number of reoperations and complications such as postoperative infections or not.
2. Evaluate the aesthetic results and the patients' experiences. For both these aims the hypothesis is that pre-treatment is in favour for the outcomes.

DETAILED DESCRIPTION:
All patients will undergo breast reconstruction with expander implant. Half of the patients will be randomized to pre-treatment with lipofilling before the reconstruction. The randomization will be carried out with block randomization. A certain person that has not met the patients has been assigned to do this.

Fat transplantation: The fat will be harvested manually with dry technique using a Coleman cannula on a 10 ml syringe. There after the syringes and fat are centrifuged at 3000 rpm for 3 minutes. Liquid fat from lysed cells and blood will be separated from the purified fat cells and discarded. The fat graft will then be injected fan-shaped in multiple layers into the subcutaneous tissues of the breast using another blunt cannula with a diameter of 1.29 mm. If necessary to obtain a volume of 100 ml fat injected the procedure will be repeated. All sessions will be performed under general anesthesia in day surgery. Three month later the patients will undergo breast reconstruction with expander prosthesis.

Those patients that are randomized to not undergo pre-treatment will undergo breast reconstruction with expander prosthesis immediately.

After the reconstruction all patients will have as many appointments as necessary for expansion with a breast nurse at our clinic. If necessary the patient will also meet the surgeon. After the month the patients have a routine doctors appointment. After 6, 12 and 24 month the patients will be followed up with objective measurements of breast symmetry and they will fill in quality of life formularies. In this study we are using the validated formulary called Breast Q and a study specific formulary. At 24 month standardized photos of the breasts will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Previously undergone mastectomy and adjuvant radiotherapy.
* Will undergo breast reconstruction with expander prosthesis.
* Mammogram and ultrasound performed maximum three month prior surgery.
* At least one year since last operation or radiotherapy.

Exclusion Criteria:

* Known breast cancer relapse
* Distant metastases except axillary
* Any contraindication for anaesthesia
* Systemic disease such as diabetes mellitus type I.
* BMI >30 (if the patients lose weight they are eligible)

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-10; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of reoperations | Two years on from reconstruction with prosthesis
Frequency of complications | Two years on from reconstruction with prosthesis

SECONDARY OUTCOMES:
Total days in hospital during fat transplantation and reconstruction with prosthesis | 4 month
  Number of days spent at the hospital for surgery including both day surgery with fat transplantation and reconstruction with prosthesis.
Number of appointments as outpatient after breast reconstruction. | Two years on from reconstruction with prosthesis
  Number of appointments with surgeon and nurse as outpatient after the reconstructive surgery is performed.
Aesthetic evaluation of the results of the breast reconstruction | Two years on from reconstruction with prosthesis
  Aesthetic outcome is evaluated by plastic surgeons through assessment of standardized photographies of the patients.
Patient reported outcome | Measured at 6, 12 and 24 month from reconstruction with prosthesis
  Breast Q is a validated questionnaire for quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Inkeri Schultz, PhD, Study Chair; Åsa Edsander-Nord, Docent, Study Chair; Marie Wickman Chantereau, Professor, Study Director
Locations (1):
- Karolinska Institutet, Department of Molecular Medicine and Surgery, Karolinska University Hospital, Department of Reconstructive Plastic Surgery, Stockholm, Sweden

REFERENCES:
- [Background] Serra-Renom JM, Munoz-Olmo JL, Serra-Mestre JM. Fat grafting in postmastectomy breast reconstruction with expanders and prostheses in patients who have received radiotherapy: formation of new subcutaneous tissue. Plast Reconstr Surg. 2010 Jan;125(1):12-18. doi: 10.1097/PRS.0b013e3181c49458. PMID 20048576
- [Background] Rigotti G, Marchi A, Galie M, Baroni G, Benati D, Krampera M, Pasini A, Sbarbati A. Clinical treatment of radiotherapy tissue damage by lipoaspirate transplant: a healing process mediated by adipose-derived adult stem cells. Plast Reconstr Surg. 2007 Apr 15;119(5):1409-1422. doi: 10.1097/01.prs.0000256047.47909.71. PMID 17415234
- [Background] Sarfati I, Ihrai T, Kaufman G, Nos C, Clough KB. Adipose-tissue grafting to the post-mastectomy irradiated chest wall: preparing the ground for implant reconstruction. J Plast Reconstr Aesthet Surg. 2011 Sep;64(9):1161-6. doi: 10.1016/j.bjps.2011.03.031. Epub 2011 Apr 22. PMID 21514910
- [Background] Mojallal A, Lequeux C, Shipkov C, Breton P, Foyatier JL, Braye F, Damour O. Improvement of skin quality after fat grafting: clinical observation and an animal study. Plast Reconstr Surg. 2009 Sep;124(3):765-774. doi: 10.1097/PRS.0b013e3181b17b8f. PMID 19730294
- See also: Swedish Breast Cancer Group. Provides national guidelines for breast cancer treatment etc. — http://www.swebcg.se/index.asp?P=Start